CLINICAL TRIAL: NCT02582073
Title: Double-blind Randomized Parallel Group Study of 3 Cumulative Doses of Grass MATA MPL Compared to Placebo and Grass MATA in Patients With Seasonal Allergic Rhinoconjunctivitis Exposed to Grass Pollen in mEECs™ Out of the Grass Pollen Season
Brief Title: Dose Selection Study of Efficacy and Safety of Different Doses of Grass MATA MPL and Grass MATA Using mEECs™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GrassMATAMPL204
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (0.5ml) (Placebo Comparator): Six 0.5ml injections of placebo consisting of L-Tyrosine, Ph. Eur 2%
  Interventions: Biological: Placebo (0.5ml)
- Placebo (1.0ml) (Placebo Comparator): Six 1.0ml injections of placebo consisting of L-Tyrosine, Ph. Eur 2%
  Interventions: Biological: Placebo (1.0ml)
- Grass MATA MPL (0.5ml) 5100SU (Experimental): Six 0.5 mL injections sequentially of placebo, placebo, 300, 800, 2000 and 2000 SU of Grass MATA with 50 µg/0.5 mL of MPL® adjuvant adsorbed to L tyrosine (2%) and 0.5% phenol (cumulative dose 5100SU).
  Interventions: Biological: Placebo (0.5ml); Biological: Grass MATA MPL (0.5ml) 5100SU
- Grass MATA MPL (1.0ml) 10200SU (Experimental): Six 1.0 mL injections sequentially of placebo, placebo, 600, 1600, 4000 and 4000 SU of Grass MATA per 1.0 mL and 50 µg/1.0 mL of MPL® adjuvant adsorbed to L tyrosine (2%) and 0.5% phenol (cumulative dose 10200 SU).
  Interventions: Biological: Placebo (1.0ml); Biological: Grass MATA MPL (1.0ml) 10200SU
- Grass MATA MPL (1.0ml) 18200SU (Experimental): Six 1.0 mL injections sequentially of placebo, 600, 1600, 4000, 4000, 4000 and 4000 SU of Grass MATA per 1.0 mL and 50 µg/1.0 mL of MPL® adjuvant adsorbed to L tyrosine (2%) and 0.5% phenol (cumulative dose 18200 SU).
  Interventions: Biological: Placebo (1.0ml); Biological: Grass MATA MPL (1.0ml) 18200SU
- Grass MATA (0.5ml) 5100SU (Active Comparator): Six 0.5ml injections sequentially of placebo, placebo, 300, 800, 2000 and 2000 SU of Grass MATA adsorbed to L tyrosine (2%) and 0.5% phenol (cumulative dose 5100SU).
  Interventions: Biological: Placebo (0.5ml); Biological: Grass MATA (0.5ml) 5100SU

INTERVENTIONS:
Biological: Placebo (0.5ml)
  Arms: Grass MATA (0.5ml) 5100SU; Grass MATA MPL (0.5ml) 5100SU; Placebo (0.5ml)
Biological: Placebo (1.0ml)
  Arms: Grass MATA MPL (1.0ml) 10200SU; Grass MATA MPL (1.0ml) 18200SU; Placebo (1.0ml)
Biological: Grass MATA MPL (0.5ml) 5100SU
  Arms: Grass MATA MPL (0.5ml) 5100SU
Biological: Grass MATA MPL (1.0ml) 10200SU
  Arms: Grass MATA MPL (1.0ml) 10200SU
Biological: Grass MATA MPL (1.0ml) 18200SU
  Arms: Grass MATA MPL (1.0ml) 18200SU
Biological: Grass MATA (0.5ml) 5100SU
  Arms: Grass MATA (0.5ml) 5100SU

SUMMARY:
There is increasing evidence that the effectiveness of allergy immunotherapy to control symptoms of rhinoconjunctivitis is related to the cumulative dose of allergen or allergoid administered during a single regimen of subcutaneous (SC) injections or of sublingual administration. The current therapeutic dose regimen for Grass MATA MPL is a course of four injections of 300, 800, 2000 and 2000 SU (Standardized Units), administered at weekly intervals (cumulative dose 5100 SU). Two new cumulative doses of the Grass MATA MPL 10200 SU and 18200 SU are being developed to compare with the current dose. The study is designed to explore the benefit/risk of increasing the cumulative allergen dose of the Grass MATA MPL immunotherapy comparing these doses with the current dose of Grass MATA MPL, Grass MATA (without MPL) and placebo.

DETAILED DESCRIPTION:
This study will be conducted outside the grass pollen season and is comprised of five periods.

* Period 1: Screening visit
* Period 2: Eligibility and baseline symptom assessments in the mobile environmental exposure chamber (mEEC™)
* Period 3: Six treatment visits, during which the study drug will be injected
* Period 4: Post-treatment efficacy assessments in the mEEC™
* Period 5: Safety follow-up

Period 1 is the screening visit (Visit 1), and will occur 3 to 28 days before Visit 2.

Period 2 includes the pre-randomization, grass pollen exposure visits, which consist of four 3 hour sessions in the mEEC™ (Visits 2, 3, 4 and 5) during which patients will be exposed to grass pollen and record nasal and non nasal symptoms using electronic diaries (electronic Patient Data Acquisition Tablet: ePDAT™) prior to entry and every 30 minutes post entry into the mEEC™. Patients will attend mEEC™ visits on consecutive days. To be eligible for randomization and proceed to Treatment (Period 3), patients must achieve the following by the final pre treatment mEEC™ (Visit 5):

* Minimum qualifying Total Symptom Score (TSS) of at least 12 out of a possible 24 on at least one exposure using ePDAT™
* Total Nasal Symptom Score (TNSS) of at least 7 out of a possible 12 using ePDAT™
* Runny nose score of at least 2 out of 3 on at least two time points.

Period 3 includes the six treatment visits (Visit 6, 7, 8, 9, 10 and 11). After each injection, patients will be kept under observation by personnel qualified to manage systemic allergic reactions at the site for at least 30 minutes. This period can be extended by the investigator in response to injection site or systemic allergic reactions. The observation will be followed up by a telephone call approximately 24 hours later.

Period 4 consists of four 3 hour sessions (Visits 12, 13, 14 and 15) in the mEEC™ during which patients will be exposed to grass pollen and record post-treatment TSS using the ePDAT™ as in Period 2.

Period 5 consists of an End of Study (EOS) safety follow-up visit (Visit 16) between 2 and 14 days after the last EEC visit. A telephone follow-up will be made at approximately 3, 6, and 12 months following the last injection with detailed enquiry with regard to expected and non-expected AEs, with special attention to New Onset Autoimmune Disorders (NOAD) and Neuro-inflammatory (NI) disease. For subjects who withdraw early, similar follow up will be done at approximately 1, 3, 6, and 12 months following the last injection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 50 years inclusive
2. Allergy to grass pollen allergen, defined by:

   1. A history of moderate to severe symptoms of seasonal allergic rhinitis and/or conjunctivitis due to grass pollen exposure that required repeated use of antihistamines, nasal steroids, and/or leukotriene modifiers for relief of symptoms, confirmed by the patient record if available.
   2. A positive skin prick test for grass pollen allergen (wheal (longest diameter) of ≥ 5 mm greater than the negative control after skin prick testing) at Visit 1.
   3. Specific IgE for grass pollen as documented by a specific IgE immunoassay, or equivalent test, with class ≥ 2 to grass pollen mix. Results from tests conducted under a generalized screening protocol within the past six months may be used and will not need to be repeated at V1 provided a copy of the test results is added to the source file.
3. Positive skin prick test to histamine (wheal (longest diameter) ≥ 3 mm greater than the negative control)
4. Negative skin prick test to the negative control (redness with wheal ≤ 2 mm is acceptable)
5. For asthmatic patients: Forced expiratory volume (FEV) in 1 second (FEV1) ≥ 80% of National Health and Nutrition Examination Surveys (NHANES) predicted, with a FEV1/Forced Vital Capacity (FVC) ratio ≥ 70%
6. Obtain the minimum qualifying symptom scores by the final pre treatment EEC visit to be enrolled into the study. Minimum qualifying TSS is at least 12 out of a possible 24 on at least one recording time, a TNSS score of at least 7 out of a possible 12 on at least one recording time, and a rhinorrhea score of at least 2 on at least two diary cards.
7. Observe the drug washout times for antihistamines, steroids etc. as specified in the protocol prior to screening (Visit 1). The use of other medications will be permitted if they are not expected to interfere with the ability of the patient to participate in the study and provided they have been on a stable regimen (i.e., the same dosage and administration) for six weeks prior to screening
8. Males or non pregnant, non lactating females who are:

   1. Post menopausal (defined as at least 12 months natural spontaneous amenorrhea or at least 6 weeks following surgical menopause, i.e. bilateral oophorectomy)
   2. Naturally or surgically sterile (hysterectomy; bilateral oophorectomy; bilateral tubal ligation with surgery at least 6 weeks prior to study initiation)
   3. Of childbearing potential - with negative urinary and serological pregnancy test and use at least one of the following contraception methods:

   i. Stable hormonal contraceptive for ≥ 90 days prior to Visit 1 and for at least 7 days after the final injection. If < 90 days prior to the study, additional use of a double barrier method until 90 days reached is required.

   ii. Placement of an intrauterine device (IUD) or intrauterine system iii. Use of barrier methods of contraception (e.g., condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository iv. Use of double barrier methods of contraception (e.g., male condom with diaphragm, male condom with cervical cap) v. Male sterilization with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate of the sole partner vi. True abstinence, when in line with the preferred and usual lifestyle of the patient; periodic abstinence, such as calendar, ovulation, symptothermal, post ovulation methods, and withdrawal are not acceptable methods of contraception.
9. Normally active and otherwise judged to be in good health on the basis of medical history, physical examination and routine laboratory tests.
10. Willing and able to give written informed consent.
11. Able to understand and comply with study instructions.
12. Willing and able to attend required study visits.

Exclusion Criteria:

1. In the presence of symptoms outside the grass pollen season coupled with a positive skin test to a perennial allergen, if as assessed by the Investigator the patient is unable to avoid the offending allergen.
2. Concurrent disease that might complicate or interfere with investigation or evaluation of the study medications or the skin prick test result, such as:

   1. Nasal polyposis
   2. Any ocular disorder (other than allergic conjunctivitis) including presumed infectious ocular disease (bacterial, fungal, viral, etc.), which could interfere with the evaluation of the study medication
   3. Rhinitis medicamentosa
   4. Documented evidence of acute or significant chronic sinusitis or upper or lower respiratory tract infection within 30 days before Visit 2 as determined by the Investigator
   5. Asthma, with the exception of mild asthma as, to lessen confounding by asthma medications. Patients taking corticosteroids for asthma at doses higher than budesonide MDI 400µg once a day or equivalent, as defined by the current GINA guideline, will be excluded.
3. Emergency room visit or admission for asthma in the 12 months prior to Visit 1 or history of a life-threatening asthma attack ever
4. Presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence
5. Presence of secondary alterations at the affected organ (i.e., emphysema, and bronchiectasis )
6. Current diagnosis of Type I diabetes. Patients with Type II diabetes will only be allowed to participate at the discretion of the Investigator
7. Autoimmune disease (e.g., of liver, kidney, lung, thyroid, nervous system, rheumatoid diseases) sarcoidosis, or NI disease (e.g., optic neuritis, multiple sclerosis or other demyelinating disease, encephalitis or encephalomyelitis, myelitis/transverse myelitis, myasthenia gravis, Guillain Barré syndrome, unexplained transitory neurological events)
8. History of cancer (excluding basal cell carcinoma) or concomitant illness (e.g., cardiovascular, pulmonary, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic, or psychiatric diseases or disorders) that, in the opinion of the Investigator, would pose a safety risk or compromise the interpretation of efficacy for this grass immunotherapy
9. Use of oral, intramuscular, intravenous corticosteroids, or potent or super-potent topical corticosteroids, from 30 days prior to screening up to Visit 16
10. Any systemic disorder that could interfere with the evaluation of the study medications
11. Presence of tattoos or other skin abnormalities in the upper arms which would prevent an accurate assessment of local skin reaction, at Investigator's discretion
12. Clinical history of allergy, hypersensitivity or intolerance to the excipients of the study medication
13. Active or quiescent tuberculous infection of the respiratory tract, untreated local or systemic fungal or bacterial or systemic viral infections (e.g., chickenpox or measles) or parasitic or ocular herpes simplex
14. Experience of nasal septal ulcers, nasal surgery or nasal trauma within 90 days of Visit 1
15. Clinical history of anaphylactic reactions to foods, insect venom, exercise, drugs or idiopathic anaphylaxis
16. Clinical history of immunodeficiency, including those who are on immunosuppressant therapy
17. Diseases with a pathogenesis interfering with the immune response and who have received medication which could influence the results of the study
18. Clinical history of recurrent idiopathic angioedema
19. Tyrosine metabolism disorders, especially tyrosinemia and alkaptonuria
20. β blocker medication, including eye drops, for any indication
21. Monoamine Oxidase Inhibitor medication
22. Unable to receive epinephrine therapy (i.e., use of epinephrine is contraindicated)
23. Clinical history of drug or alcohol abuse which would, at the Investigator's discretion, interfere with the patient's participation in the study
24. Clinical history, or evidence, of nasolacrimal drainage system malfunction
25. Any clinically significant abnormal laboratory value (as determined by the Investigator) at Visit 1
26. Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol or people considered as vulnerable or institutionalized
27. Have undergone specific immunotherapy with comparable allergen extracts. An exception will be allowed if prior immunotherapy with comparable allergen was successful, symptoms reappeared sometime after stopping the immunotherapy, and the immunotherapy was completed ≥ 3 years before Visit 1
28. Treatment with a preparation containing MPL® within 6 months prior to Visit 1
29. Participation in a clinical research study with an investigational medicinal product within 4 weeks of Visit 1 or concomitantly with this study, including the safety follow-up period up to 12 months following the last injection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Actual)
Dates: Start 2015-11-07 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Post-treatment TSS | 21-28 days after the last injection
  The primary efficacy endpoint will be the mean average of the last three TSS measurements recorded in each of the four post-treatment Visits 12 15. TSS will be measured during the four post-treatment mEEC™ sessions conducted on consecutive days 12-15, and is defined as the sum of individual NSS (rhinorrhea, congestion, sneezing and itchiness) and NNSS (itchy/gritty eyes, tearing/watery eyes, red/burning eyes and ear/palate itching).

SECONDARY OUTCOMES:
Frequency of local adverse events (AEs) | A Local AE is located at the injection site of study medication, occurring within 24 hours after the injection.
  A Local AE is located at the injection site of study medication, occurring within 24 hours after the injection.
Frequency of systemic adverse events (AEs) | 24 hours following each injection
  A Systemic AE is allergic signs and symptoms (e.g., conjunctivitis, rhinitis, cough and generalized urticaria including anaphylaxis) associated with the injection of study medication, occurring within 24 hours after the injection.
Frequency of other AEs | Up to 1 year following injections
  All post-treatment AEs that do not fall into local or systemic AEs
Frequency of AEs of special interest (AESI) | Up to 1 year following injections
  AESI includes New Onset Autoimmune Disorders and Neuro-inflammatory events.
Safety laboratory values | Up to 12 weeks
  Change in serum chemistry and haematology from baseline to Visit 16
Specific IgE | Up to 12 weeks
  Change in grass specific IgE from baseline to Visit 16

CONTACTS AND LOCATIONS:
Overall Officials: Tim Higenbottam, DSc MD FRCP, Study Director — Allergy Therapeutics
Locations (1):
- Inflamax Research Inc., Neptune City, New Jersey, United States